CLINICAL TRIAL: NCT02159287
Title: Study of the Efficacy, Safety and Tolerability of Low Molecular Weight Heparin vs. Unfractionated Heparin as Bridging Therapy in Patients With Embolic Stroke Due to Atrial Fibrillation
Brief Title: Study of the Efficacy, Safety and Tolerability of Low Molecular Weight Heparin vs. Unfractionated Heparin in Stroke
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Afshin Borhani-Haghighi, Associate Professor of Neurology Shiraz University of Medical Sciences, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 92-01-01-5667
Record Dates: First submitted 2014-01-20; First posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Embolic Stroke
Keywords: ischemic stroke; atrial fibrillation; bridging therapy
MeSH Terms: conditions — Embolic Stroke; Ischemic Stroke; Atrial Fibrillation | interventions — Enoxaparin; Heparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low molecular-weight heparin (Experimental): these patients will receive 1 mg of enoxaparin (clexane) per kilogram of body weight subcutaneous every 12 hour with warfarin 5mg QD and both drugs will be continued until the target INR level (2.5) is reached then clexane will be discontinued.
  Interventions: Drug: Enoxaparin
- unfractionated heparin (Active Comparator): This group will receive continuous intravenous unfractionated heparin sodium infusion 1000 unit per hour initially and then the dose will be adjusted to maintain a therapeutic aPTT level (two times to baseline) then warfarin will be started (5 mg QD).
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Enoxaparin — 1 mg of enoxaparin per kilogram of body weight subcutaneous every 12 hour
  Other Names: clexane (Clexane, Sanofi, Paris)
  Arms: Low molecular-weight heparin
Drug: Heparin — 1000 unit per hour continuous intravenous infusion of heparin sodium
  Other Names: Heparin Sodium (Alborz Darou,Tehran)
  Arms: unfractionated heparin

SUMMARY:
Patients with Atrial fibrillation (AF) make a unique group of ischemic stroke, mostly caused by emboli from the left atrial appendage. Oral anticoagulation (Warfarin) is recommended for prevention of recurrent embolic stroke but it takes several days to reach a therapeutic international normalized ratio (INR : 2.5) so bridging therapy with a short acting intravenous anticoagulant is recommended until therapeutic INR level is reached. A common strategy is to use intravenous unfractionated heparin (UFH) until a standard activated partial thromboplastin time (aPTT) is reached and then initiating warfarin. Another strategy is to use subcutaneous (SQ) injection of a low-molecular-weight heparin (LMWH) eg. Enoxaparin.

The investigators will compare LMWH and UFH, focusing on risk of new stroke and mortality rate.

METHOD: This study is randomized controlled trial that will be performed in 80 patients ages between 18 and 75 with confirmed acute ischemic stroke purely due to AF who will be hospitalized in Shiraz Medical University affiliated teaching hospitals. Patients will be randomly assigned in two groups. A brain CT will be done to confirm the absence of intracranial hemorrhage and to assess the size of cerebral ischemia.

First group will receive 1 mg of enoxaparin (Clexane, Sanofi, Paris) per kilogram of body weight SQ every 12 hour with warfarin 5mg orally everyday and both drugs will be continued until the target INR level (2.5) is reached then clexane will be discontinued.

The second group will receive continuous UFH infusion 1000 unit per hour and then the dose will be adjusted to maintain a therapeutic aPTT (two times to baseline) level then warfarin will be started (5 mg everyday).

The investigators will follow patients in both groups until target INR will be achieved (2.5) and after that clexane and UFH will be discontinued. Adverse events will be assessed in both groups for three months.

Data will be analyzed with Statistical Package for the Social Sciences (SPSS) version 15 and Chi-square statistics.

Main outcome of our study will be evaluation of new stroke, mortality, central nervous system (CNS) hemorrhage, major bleeding, drop out and other unwanted side effects in first week and three months after stroke.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of acute ischemic stroke purely due to AF
* AF confirmed by ECG or 24 hour holter monitoring
* patients who need initiation of anticoagulation for prevention of recurrent stroke

Exclusion Criteria:

* ages less than 18 or more than 75
* no cooperation
* CNS hemorrhage
* major bleeding
* infarction size of more than one third of middle cerebral artery territory
* National Institutes of Health Stroke Scale (NIHSS) more than 20
* hypersensitivity to IV UFH or LMWH
* no informed consent
* other causes for stroke except AF
* pregnancy
* breast feeding
* uncontrolled hypertension (BP more than 220/120)
* renal, hepatic, respiratory or cardiac failure
* myocardial infarction
* infectious endocarditis
* coma
* vasculitis
* dissection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-02 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
mortality | up to the 3 months of follow-up
  all death cases are included but only mortality due to cerebrovascular accident are considered.
ischemic stroke | up to the 3 months of follow-up
  Ischemic strokes are those that are caused by interruption of the blood supply
hemorrhagic stroke | up to the 3 months of follow-up
  hemorrhagic strokes are the ones which result from rupture of a blood vessel or an abnormal vascular structure.

SECONDARY OUTCOMES:
symptomatic CNS hemorrhage | up to the 3 months of follow-up
  Intracranial bleeding occurs when a blood vessel within the skull is ruptured or leaks that causes neurological symptoms. It can result from nontraumatic causes as occurs in hemorrhagic stroke such as a ruptured aneurysm. Anticoagulant therapy can heighten the risk that an intracranial hemorrhage will occur.
Non-CNS hemorrhage | up to the 3 months of follow-up
  any bleeding of other sites of body except CNS.
asymptomatic CNS_hemorrhage | up to the 3 months of follow-up
  Intracranial bleeding occurs when a blood vessel within the skull is ruptured or leaks that will not cause neurological symptoms. It can result from nontraumatic causes as occurs in hemorrhagic stroke such as a ruptured aneurysm. Anticoagulant therapy can heighten the risk that an intracranial hemorrhage will occur.
time to reach target INR | average time 7 to 10 days (it is variable between individuals)
  the therapeutic INR level for patients on warfarin therapy is between 2.0 to 3.0.
tolerability of drugs | participants will be followed for the duration of hospital stay, an expected average of 1 week
  tolerability is how a patient can tolerate heparin and LMWH in terms of side effect and route of administration.

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Borhani Haghighi, Associate professor, Principal Investigator — Shiraz University of medical sciences, department of neurology; Farnia Feiz, medical student, Study Chair — Shiraz University of Medical Sciences; Reyhane Sedghi, medical student, Study Chair — Shiraz University of Medical Sciences
Locations (2):
- Iran (2):
  - Nemazi hospital, Shiraz, Fars
  - Faghihi hospital, Shiraz, Fars

REFERENCES:
- [Background] Shahpouri MM, Mousavi S, Khorvash F, Mousavi SM, Hoseini T. Anticoagulant therapy for ischemic stroke: A review of literature. J Res Med Sci. 2012 Apr;17(4):396-401. PMID 23267405
- [Background] Kase CS, Albers GW, Bladin C, Fieschi C, Gabbai AA, O'Riordan W, Pineo GF; PREVAIL Investigators. Neurological outcomes in patients with ischemic stroke receiving enoxaparin or heparin for venous thromboembolism prophylaxis: subanalysis of the Prevention of VTE after Acute Ischemic Stroke with LMWH (PREVAIL) study. Stroke. 2009 Nov;40(11):3532-40. doi: 10.1161/STROKEAHA.109.555003. Epub 2009 Aug 20. PMID 19696423
- [Background] Algra A, de Schryver EL, van Gijn J, Kappelle LJ, Koudstaal PJ. Oral anticoagulants versus antiplatelet therapy for preventing further vascular events after transient ischaemic attack or minor stroke of presumed arterial origin. Cochrane Database Syst Rev. 2001;(4):CD001342. doi: 10.1002/14651858.CD001342. PMID 11687110
- [Background] Saxena R, Lewis S, Berge E, Sandercock PA, Koudstaal PJ. Risk of early death and recurrent stroke and effect of heparin in 3169 patients with acute ischemic stroke and atrial fibrillation in the International Stroke Trial. Stroke. 2001 Oct;32(10):2333-7. doi: 10.1161/hs1001.097093. PMID 11588322
- [Background] Hallevi H, Albright KC, Martin-Schild S, Barreto AD, Savitz SI, Escobar MA, Gonzales NR, Noser EA, Illoh K, Grotta JC. Anticoagulation after cardioembolic stroke: to bridge or not to bridge? Arch Neurol. 2008 Sep;65(9):1169-73. doi: 10.1001/archneur.65.9.noc70105. Epub 2008 Jul 14. PMID 18625852
- [Background] Guyatt GH, Akl EA, Crowther M, Gutterman DD, Schuunemann HJ; American College of Chest Physicians Antithrombotic Therapy and Prevention of Thrombosis Panel. Executive summary: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):7S-47S. doi: 10.1378/chest.1412S3. No abstract available. PMID 22315257
- [Background] Fahimi F, Baniasadi S, Behzadnia N. Enoxaparin Utilization Evaluation: An Observational Prospective Study in Medical Inpatients. Iranian Journal of Pharmaceutical Research 2008;7 (1):77-82.
- [Background] Kalafut MA, Gandhi R, Kidwell CS, Saver JL. Safety and cost of low-molecular-weight heparin as bridging anticoagulant therapy in subacute cerebral ischemia. Stroke. 2000 Nov;31(11):2563-8. doi: 10.1161/01.str.31.11.2563. PMID 11062276
- [Background] Adams HP Jr, del Zoppo G, Alberts MJ, Bhatt DL, Brass L, Furlan A, Grubb RL, Higashida RT, Jauch EC, Kidwell C, Lyden PD, Morgenstern LB, Qureshi AI, Rosenwasser RH, Scott PA, Wijdicks EF; American Heart Association; American Stroke Association Stroke Council; Clinical Cardiology Council; Cardiovascular Radiology and Intervention Council; Atherosclerotic Peripheral Vascular Disease and Quality of Care Outcomes in Research Interdisciplinary Working Groups. Guidelines for the early management of adults with ischemic stroke: a guideline from the American Heart Association/American Stroke Association Stroke Council, Clinical Cardiology Council, Cardiovascular Radiology and Intervention Council, and the Atherosclerotic Peripheral Vascular Disease and Quality of Care Outcomes in Research Interdisciplinary Working Groups: the American Academy of Neurology affirms the value of this guideline as an educational tool for neurologists. Stroke. 2007 May;38(5):1655-711. doi: 10.1161/STROKEAHA.107.181486. Epub 2007 Apr 12. PMID 17431204
- [Background] Cohen M, Demers C, Gurfinkel EP, Turpie AG, Fromell GJ, Goodman S, Langer A, Califf RM, Fox KA, Premmereur J, Bigonzi F. A comparison of low-molecular-weight heparin with unfractionated heparin for unstable coronary artery disease. Efficacy and Safety of Subcutaneous Enoxaparin in Non-Q-Wave Coronary Events Study Group. N Engl J Med. 1997 Aug 14;337(7):447-52. doi: 10.1056/NEJM199708143370702. PMID 9250846
- [Background] Burak CR, Bowen MD, Barron TF. The use of enoxaparin in children with acute, nonhemorrhagic ischemic stroke. Pediatr Neurol. 2003 Oct;29(4):295-8. doi: 10.1016/s0887-8994(03)00270-4. PMID 14643390